CLINICAL TRIAL: NCT05708339
Title: Adaptation of Conventional Versus Virtually Fabricated Ear Prosthesis in Patients With Auricular Defects: a Randomized Controlled Trial.
Brief Title: Adaptation of Conventional Versus Virtually Fabricated Ear Prosthesis in Patients With Auricular Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Elmougi (Other)
Responsible Party: Sponsor-Investigator, Fatima Elmougi, Doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19115
Record Dates: First submitted 2022-12-29; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Ear Deformity External

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventionally fabricated ear prosthesis (Active Comparator)
  Interventions: Other: conventionally fabricated ear prosthesis
- virtually fabricated ear prosthesis (Experimental)
  Interventions: Other: virtually fabricated ear prosthesis

INTERVENTIONS:
Other: virtually fabricated ear prosthesis — virtually designed ear prosthesis
  Arms: virtually fabricated ear prosthesis
Other: conventionally fabricated ear prosthesis — conventionally fabricated ear prosthesis
  Arms: conventionally fabricated ear prosthesis

SUMMARY:
: patients were recruited for auricular prosthetic reconstruction. Preoperative data was collected including personal and medical history, plain photographs and CT scans. Pre-operative prosthetic and implant planning were carried out. Three endosseous implants were placed in a two-stage surgical technique. Patients were assigned into two groups with allocation ratio 1:1. In control group, Implant level impression was recorded, and a stone model of the defect was cast. waxing up of the ear was done on the stone cast followed by flasking, wax elimination, packing of heat cured acrylic resin and curing. In intervention group, CT scanning was done to the full head and optical scanning was done to the defect site with scan bodies screwed to the implants. Using Exocad software a model of the defect site with implant analogues and ear model with abutment extensions were planned and printed using SLA printing technology. A placement jig was done for ear models of both groups and adaptation was measured on the patient using silicon replica technique. The silicone replica was sectioned and the gap, represented in light consistency polyvinyl siloxane impression material was measured using digital microscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missing or severely deformed ears.
* Patients with failed autogenous reconstruction.
* Compliant and cooperative patients.
* Patients committed to maintain the prosthesis.
* Patients willing to attend the follow up appointments.

Exclusion Criteria:

* Patients undergoing radiotherapy or chemotherapy treatment.
* Patients taking corticosteroids or bisphosphonates.
* Patients with contraindications for CT scanning.
* Patients with any debilitating medical condition.
* Patients with any type of psychosomatic disorder.
* Patients allergic to any of the materials used.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Prosthesis adaptation using Silicon replica measuring technique. | Day 1
  measuring gap between prosthesis and defect

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No